CLINICAL TRIAL: NCT06226623
Title: Effects of Coconut Consumption on Body Composition in Healthy Adult Individuals: a Randomized Controlled Study
Brief Title: Effect of Coconut Consumption on Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Betul Uner, Lecturer, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: There is no sponsor support.
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Body Composition
Keywords: Coconut, Body Composition, Healthy Eating

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled study. The research was single-centered and was carried out with the academic, administrative and other personnel of Muğla Sıtkı Koçman University Faculty of Health Sciences. A list of all faculty members was created by the researchers. Randomization was made to the experimental and control groups in a 1:1 ratio using the sealed envelope selection method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants were given 4-week healthy nutrition training. Participants' basal metabolic rates were calculated according to gender and body weight (kg) using the Schofield equation. The appropriate equation for each participant's age was used. The daily energy requirement of the participants was calculated by adding an activity factor of 1.3 to the calculated basal metabolic rate. A healthy nutrition program was prepared according to the calculated daily energy needs of the participants. While preparing this program, WHO and Turkey-Specific Healthy Nutrition Guide (TÜBER) were used. In the individual healthy nutrition program, 55% carbohydrates, 15% protein and 30% fat macronutrients were provided. Total cholesterol of the nutrition program was kept at 300 mg and below. The intervention group was asked to consume 50 g of fresh coconut daily in addition to the healthy nutrition program.
  Interventions: Dietary Supplement: Coconut
- Control (No Intervention): Participants were given 4-week healthy nutrition training. Participants' basal metabolic rates were calculated according to gender and body weight (kg) using the Schofield equation. The appropriate equation for each participant's age was used. The daily energy requirement of the participants was calculated by adding an activity factor of 1.3 to the calculated basal metabolic rate. A healthy nutrition program was prepared according to the calculated daily energy needs of the participants. While preparing this program, WHO and Turkey-Specific Healthy Nutrition Guide (TÜBER) were used. In the individual healthy nutrition program, 55% carbohydrates, 15% protein and 30% fat macronutrients were provided. Total cholesterol of the nutrition program was kept at 300 mg and below. The control group was given only a healthy nutrition program.

INTERVENTIONS:
Dietary Supplement: Coconut — Participants in the intervention group, unlike participants in the control group, were asked to consume 50 g of fresh coconut daily for four weeks.
  Arms: Intervention

SUMMARY:
This research is a randomized controlled study. The aim of the study is to investigate the effects of coconut on body composition, compare our results with other studies in the literature and contribute to the field.

The research was single-centered and was carried out with the academic, administrative and other personnel of Muğla Sıtkı Koçman University Faculty of Health Sciences. Volunteer, healthy adults between the ages of 18-65, without any physical disability or uncontrolled chronic systemic disease or problems with reading and comprehension, were included in the study, regardless of gender. Individuals who were following an existing diet program, having a history of pregnancy and cancer, having undergone acute abdominal surgery, or having unstable conditions due to cardiovascular and endocrine systems were not included in the study. Participants who did not attend the four-week healthy nutrition training were excluded from the study.

A list of all staff members at the faculty was created. The population of the research consists of 74 personnel. Randomization was made to the experimental and control groups by the sealed envelope selection method.

All participants were given 4 weeks of healthy nutrition training. The amount of energy required by the participants was calculated. A healthy nutrition program was prepared according to the calculated daily energy needs of the participants. The control group was given only a healthy nutrition program. The intervention group was asked to consume 50 g of fresh coconut daily in addition to the healthy nutrition program. Participants' compliance with the healthy nutrition program and coconut consumption was high.

Anthropometric measurements of the volunteer individuals participating in the study were taken before and after the intervention. To determine the body composition of individuals, a bioelectric impedance analyzer was used, a portable height meter was used to measure height, and waist circumference was measured using a standard non-stretchable tape measure. Body Mass Index (BMI) was calculated.

DETAILED DESCRIPTION:
This research is a randomized controlled study. The research was single-centered and was carried out with the academic, administrative and other personnel of Muğla Sıtkı Koçman University Faculty of Health Sciences. Participants who agreed to participate in this study and were deemed eligible were given detailed information about the research and then an informed consent form was presented in writing and signed. The study was conducted within the framework of the standards and ethical criteria in the Declaration of Helsinki and was approved by Bahçeşehir University Clinical Research Ethics Committee (2018-05/05). This research was written according to CONSORT criteria.

The study was conducted between January and July 2018. Volunteer, healthy adults between the ages of 18-65, without any physical disability or uncontrolled chronic systemic disease or problems with reading and comprehension, were included in the study, regardless of gender. Individuals who were following an existing diet program, having a history of pregnancy and cancer, having undergone acute abdominal surgery, or having unstable conditions due to cardiovascular and endocrine systems were not included in the study. Participants who did not attend the four-week healthy nutrition training were excluded from the study.

A list of all faculty members was created by the researchers. Randomization was made to the experimental and control groups in a 1:1 ratio using the sealed envelope selection method. Data was collected between April and May 2018.

Power analysis was used to calculate the sample size of this study. Since G Power power analysis was performed with a 95% confidence interval and an effect size of 0.8, it was found that 20 participants per group should be included in the study. The population of the research includes 74 personnel. In this study, the target for the number of samples is to reach the universe. However, the sample of the study consisted of 62 personnel who met the inclusion criteria and agreed to participate in the study voluntarily.

All participants were given 4 weeks of healthy nutrition training. Participants' basal metabolic rates were calculated according to gender and body weight (kg) using the Schofield equation. The equation appropriate for each participant's age was used. The daily energy requirement of the participants was calculated by adding an activity factor of 1.3 to the calculated basal metabolic rate. A healthy nutrition program was prepared according to the calculated daily energy needs of the participants. While preparing this program, WHO and Turkey-Specific Healthy Nutrition Guide (TÜBER) were used. In the individual healthy nutrition program, 55% carbohydrates, 15% protein and 30% fat macronutrients are provided. Total cholesterol in the nutrition program was kept at 300 mg and below. The control group was given only a healthy nutrition program. The intervention group was asked to consume 50 g of fresh coconut daily in addition to the healthy nutrition program. Coconuts were regularly provided to the participants as a whole fruit by the researchers.

The intervention program lasted 4 weeks. Face-to-face interviews lasting approximately 30 minutes were held with all participants every week. With these interviews, the compliance of the intervention and control groups with the healthy nutrition program and coconut consumption was evaluated. Participants' compliance with the healthy nutrition program and coconut consumption was high.

Anthropometric measurements of the volunteer individuals participating in the study were taken before and after the intervention. Tanita brand SC 330 model bioelectric impedance analyzer, which is frequently used in the literature, was preferred to determine the body composition of individuals. In addition, height was measured using a portable height meter that can measure between 14-200 cm, and waist circumference was measured using a standard rigid tape measure. Body Mass Index (BMI) was calculated.

Tanita brand SC 330 model Bioelectrical Impedance Analysis (BIA) device, which has a measurement accuracy of 0.1 kg, was used to determine body composition. With this device, the body weights of individuals were measured, and a document calculating muscle and fat masses, fat percentages and basal metabolic rates was obtained thanks to the 50 kHz electric current it sent to the body. BIA is one of the anthropometric measurement methods. BIA analysis, which is a quick and non-invasive method, is based on the principle that the resistance of fat tissue to the electrical current passed through the body is different from other tissues; It is a measurement method with high validity and reliability used to objectively calculate body fat mass. In order to obtain the most accurate results with BIA measurements, individuals should be measured with bare and dry feet three hours after getting up from bed, twelve hours after going to the toilet, twelve hours after exercising, approximately three hours after food consumption and excessive fluid intake, and before bathing, sauna and swimming.

The height of the volunteers was measured barefoot using a portable height meter that can measure between 14 and 200 cm on the Frankfort plane with an accuracy of 0.1 cm.

Waist circumference was measured at the midpoint between the last rib and the iliac bone with the help of a rigid tape measure.

Statistical Package for Social Sciences (SPSS), version 22.0 computer package program for Windows, was used for statistical analysis. Statistical data are expressed as mean ± standard deviation (X±SD), median or percentage (%). Whether the data showed normal distribution was evaluated with the Kolmogorov-Smirnov test. The significance of the changes in body weight, fat mass and percentage, waist circumference measurements and BMI values within the groups was examined using the Wilcoxon T test. The intergroup significance of the change in body composition of the individuals participating in the study was determined by the Mann Whitney U test. In statistical analysis, the significance value within and between groups was taken as p<0.05, and the difference between groups was taken as p<0.025.

ELIGIBILITY:
Inclusion Criteria:

* Without physical disability
* No problems with reading and comprehension
* Those who do not have an existing diet program,
* Non pregnant
* Not having cancer,
* Those who have not had acute abdominal surgery
* Without unstable conditions originating from the cardiovascular and endocrine systems
* Those who completed the four-week healthy nutrition training
* Voluntary based
* Healthy adults

Exclusion Criteria:

* Physically disabled
* Having problems with reading and comprehension
* Have an existing diet program
* Pregnant
* Suffering from cancer
* Those who have had acute abdominal surgery
* Unstable condition originating from the cardiovascular and endocrine systems
* Those who did not complete the four-week healthy nutrition training
* Those who do not want to participate in the study
* Adults who are not healthy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Body Composition | Anthropometric measurements of the participants were taken before and after the intervention. Anthropometric measurements were made 5 days before the intervention and 5 days after the intervention, for a total of 10 days.
  Height was measured with a portable height meter, weight, body fat percentage, and body fat mass were determined with a BIA device, and waist circumference was determined with a rigid tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Uner Yilmaz, Lecturer, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Mugla sitki Kocman University, Muğla, Mentese, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No